CLINICAL TRIAL: NCT03540446
Title: To Prove the Effectiveness of PENS Therapy With Peripheral Neuropathy
Brief Title: First Relief Treatment for Peripheral Neuropathy
Acronym: FRT-PN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FRT-PN-18
Record Dates: First submitted 2018-04-24; First posted 2018-05-30 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Neuropathy
Keywords: First Relief; Diebetes; Pheripheral Neuropathy; Pain Releif
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard stimulation (Experimental): Group A will be treated with First Relief Treatment at standard stimulation.
  Interventions: Device: First Relief Treatment
- sweep stimulation (Experimental): Group B will be treated with First Relief Treatment at sweep stimulation.
  Interventions: Device: First Relief Treatment
- Placebo (Experimental): Group C will be treated with First Relief Treatment, receiving a placebo.(dummy device with no electrical stimulation)
  Interventions: Device: First Relief Treatment

INTERVENTIONS:
Device: First Relief Treatment — To prove the effectiveness of Percutaneous Electrical Neuro-stimulation therapy for the treatment of conditions associated with peripheral neuropathy, in a double-blind environment.

SUMMARY:
To prove the effectiveness of Percutaneous Electrical Neuro-stimulation therapy for the treatment of conditions associated with peripheral neuropathy, in a double-blind environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Neuropathy pain

Exclusion Criteria:

* Patient with inbuilt pacemakers or any other devices which allows current into the body, pregnant ladies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of Neuropathy pain | According to the patients condition and other factors expected to reduce pain in 4th week of the treatment
  This treatments effective outcome will be, "Percutaneous Electrical Nerve Stimulation therapy will have the ability to reduce the pain and other conditions regarding peripheral neuropathy" which can be verified through "Biothesiometer" parameters.

SECONDARY OUTCOMES:
Check for delay of Re-occurrence of pain within a short time | 90 Days
  After the treatment of 4th week the pain will be reduced and the treatment is continued for other 3 weeks where the booster dose is applied for the assurance of delay of pain which is evaluated manually by the medical personals after 90 days of booster dose treatment

OTHER OUTCOMES:
Complete reduction of conditions associated with peripheral neuropathy | 7 weeks
  After the overall treatment has been completed the conditions associated with peripheral neuropathy will be completely reduced and the occurrence of the pain will be stopped which can be verified and evaluated through "Biothesiometer" parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gurunath, Ph.D, Study Director — Jeevak hospital
Locations (1):
- Clinic, Warangal, Telangana, India

IPD SHARING:
Plan to Share IPD: No